CLINICAL TRIAL: NCT04886258
Title: A Randomized, Two-arm, Placebo-controlled, Participant and Investigator-blinded Study Investigating the Efficacy, Safety and Tolerability of DFV890 in Patients With Symptomatic Knee Osteoarthritis
Brief Title: Study of Efficacy, Safety and Tolerability of DFV890 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDFV890B12201; 2020-006104-17 (EudraCT Number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Knee Osteoarthritis
Keywords: Osteoarthritis; Knee osteoarthritis; DFV890; Adult; NLRP3 inhibitor; Inflammasome inhibition
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFV890 (Experimental): DFV890 was administered orally twice per day, 10 mg during 2 weeks and 25 mg during the next 10 weeks.
  Interventions: Drug: DFV890
- Placebo (Placebo Comparator): Matching Placebo was administered orally twice per day during 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFV890 — DFV890 was administered orally twice per day, 10 mg during 2 weeks and 25 mg during the next 10 weeks.
  Arms: DFV890
Drug: Placebo — Matching Placebo was administered orally twice per day during 12 weeks.
  Arms: Placebo

SUMMARY:
This was a double-blinded, two-arm, phase 2a study to assess efficacy, safety and tolerability of DFV890 in participants with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
The purpose of the Phase 2a proof of concept study was to evaluate the safety and tolerability of DFV890 in participants with symptomatic knee OA, and to determine the efficacy of DFV890 in reducing knee pain as evidenced by change in KOOS (knee injury and osteoarthritis outcome score). The study had a screening period up to 45 days, a treatment period of 12 weeks and a 4-week follow-up period. At most, the study duration was 21 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants >= 50 and <= 80 years old on the day of Informed Consent signature.
* Participants must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 35 kg/m2 at screening. BMI = Body weight (kg) / [Height (m)]2
* High sensitivity C-reactive protein (hsCRP) >=1.8 mg/L at screening
* Symptomatic OA with pain (corresponding to Numeric Rating Scale [NRS] 5-9, inclusive) in the target knee for the majority of days in the last 3 months prior to screening
* KOOS pain sub-scale score <= 60 in index knee at screening and baseline
* Radiographic disease: K&L grade 2 or 3 knee osteoarthritis in the target knee, confirmed by X-ray at screening.
* Active synovial inflammation at screening (defined a summary score of ≥7 with at least one region scoring 2) on contrast enhanced MRI (CE-MRI) of the whole knee for synovitis detection from 11 sites.

Key Exclusion Criteria:

* Total WBC count < 3,000/µL, absolute peripheral blood neutrophil count (ANC) < 1,000/µL, hemoglobin < 8.5 g/dL (85 g/L) or platelet count < 100,000/µL at Screening
* Known autoimmune disease with inflammatory arthritis (including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus), crystal-induced arthritis (gout, pseudogout associated arthritis), active acute or chronic infection or past infection of the knee joint, Lyme disease involving the knee, reactive arthritis, systemic cartilage disorders, moderate to severe fibromyalgia (widespread pain index, WPI, >4 out of 19), or a known systemic connective tissue disease
* Any known active infections, including skin or knee infections or infections that may compromise the immune system, such as HIV or chronic hepatitis B or C infection. COVID-19 specific: PCR or antigen test against COVID-19 is mandatory where required by the local Health Authority and/or by local regulation, e.g. in Germany.
* Use of prohibited medications: any local i.a. treatment into the knee, including but not restricted to viscosupplementation and corticosteroids within 12 weeks prior to Day 1; long-term treatment (>14 days) with oral corticosteroids >5 mg/day within 4 weeks prior to Day 1; oral glucosamine, chondroitin sulfate, or any nutraceutical with potential activity on cartilage repairfrom screening 1; systemic Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), selective Cyclooxygenase-2 (COX- 2) inhibitors or other non-opioid analgesics not defined as basic pain medication within 5 half-lives from PRO assessments; any other immunomodulatory drugs or treatment which cannot be discontinued or switched to a different medication within 28 days or 5 half-lives of screening (whichever is longer if required by local regulations), or until the expected PD effect has returned to baseline.
* Moderate to severe pain in the contralateral knee for the majority of days in the last 3 months prior to Screening, as per patient judgment.
* Severe malalignment greater than 7.5 degrees in the target knee (either varus or valgus), measured using x-ray at Screening.

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (7):
  - ARENSIA Explor Med Res Clinic, Phoenix, Arizona
  - TriWest Reserach Associates, El Cajon, California
  - Skylight Health Res Inc Color Spr, Colorado Springs, Colorado
  - IRIS Research and Development, Plantation, Florida
  - Conquest Research, Winter Park, Florida
  - Ctr for Adv Research and Education, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Miguel, Tucumán Province
  - Novartis Investigative Site, San Miguel de Tucumán
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Germany (4):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
- Hungary (4):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Veszprém
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Bucharest
- Slovakia (2):
  - Novartis Investigative Site, Nové Mesto nad Váhom
  - Novartis Investigative Site, Piešťany
- Spain (4):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 32 investigative sites in 8 countries.
Pre-assignment Details: The study consisted of a screening period up to 45 days.
Period: Overall Study
Arm/Group | DFV890 | Placebo
Started | 58 | 57
Completed | 52 | 54
Not Completed | 6 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFV890 | Placebo | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.00) | 64.3 (7.32) | 64.1 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 13 | 9 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 1 | 3 | 4
  White | 57 | 51 | 108
  Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the pain frequency/severity during functional activities consisting of 9 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no pain and 0 indicating extreme pain) is calculated for each subscale. Change from baseline in KOOS pain score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 12
Population: Full analysis set: All randomized participants that have received any study drug and had a valid measurement at the respective time-point. Based on a primary estimand framework.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 45 | 41
score on scale | 21.7 (2.52) | 16.7 (2.61)
Statistical Analysis 1: Comparison: DFV890 vs Placebo; Test type: Other; p = 0.0872, Mixed effects model for repeated measure; Mean Difference (Net) = 4.9806, 95% CI 2-sided [-2.2 to 12.2], Standard Error of Mean 3.6408

2. Secondary Outcome: Change From Baseline in Synovitis Activity Level Measured From Ktrans by Dynamic Contrast Enhanced MRI (DCE-MRI)
Description: Magnetic resonance images (MRI) were obtained from the target knee with dynamic contrast enhancement (DCE) to visualize and quantify changes in k-trans as a marker of the activity of synovial inflammation. In dynamic contrast-enhanced MRI, ktrans is a parameter that reflects how quickly contrast agent moves from blood vessels into the surrounding tissue, capturing both blood flow and vascular permeability. In synovitis, inflamed synovial tissue shows increased perfusion and leaky microvasculature, so higher k-trans values are interpreted as indicating more active synovial inflammation. Change from baseline in synovitis activity level measured from ktrans was analyzed to compare treatment groups. The model included treatment as fixed effect and baseline as continuous covariate. Ktrans is a marker of synovial inflammation in relation to vascularity permeability.
Time Frame: Baseline, Week 12
Population: Full analysis set: All randomized participants that have received any study drug and had a valid measurement at the respective time-point. Based on a secondary estimand framework.
Measure: Least Squares Mean (Standard Error); unit: min^-1
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 39 | 35
min^-1 | -0.0029 (0.0013) | -0.0003 (0.0014)

3. Secondary Outcome: Change From Baseline in Serum High Sensitivity C-reactive Protein (hsCRP) Level
Description: HsCRP is a protein produced by the liver in response to inflammation in the body, such as from an infection, injury, or chronic inflammatory conditions. HsCRP was used to assess the effect of DFV890 compared to placebo on systemic inflammatory status.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: Full analysis set: All randomized participants that have received any study drug and had a valid measurement at the respective time-point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 56 | 57
mg/L
  Week 2 | -1.753 (3.3198) | 0.486 (2.8528)
  Week 4: number analyzed (Participants) | 53 | 56
  Week 4 | -1.783 (3.9239) | 0.541 (4.6472)
  Week 8: number analyzed (Participants) | 53 | 56
  Week 8 | -1.953 (2.3093) | -0.045 (2.1858)
  Week 12: number analyzed (Participants) | 51 | 55
  Week 12 | -0.855 (7.7378) | 1.119 (5.0495)

4. Secondary Outcome: Change From Baseline in Absolute Neutrophil Counts (ANC)
Description: ANC measures the number of neutrophils, a type of white blood cell crucial for fighting infection, in a blood sample. ANC was used to judge target engagement of DFV890.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: neutrophils*10^9/L
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 52 | 56
neutrophils*10^9/L
  Week 2 | -0.981 (1.4694) | -0.221 (0.7925)
  Week 4: number analyzed (Participants) | 51 | 52
  Week 4 | -0.980 (1.4698) | -0.054 (0.8272)
  Week 8: number analyzed (Participants) | 51 | 55
  Week 8 | -1.045 (1.2502) | -0.056 (1.1135)
  Week 12: number analyzed (Participants) | 50 | 51
  Week 12 | -1.030 (1.0915) | -0.167 (0.8977)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of DFV890
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. DFV890 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8). DFV890 was determined by a validated LC-MS/MS method; the lower limit of quantification (LLOQ) is 1 ng/mL.
Time Frame: Week 2 and Week 12: pre-dose, 1h, 3h, 5h, 8h
Population: The Pharmacokinetic (PK) analysis set included all participants with at least 1 available valid (i.e., not flagged for exclusion) PK concentration measurement, who received DFV890 and with no protocol deviations that impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DFV890
Number analyzed (Participants) | 52
ng/mL
  Week 2 | 1550 (603)
  Week 12: number analyzed (Participants) | 50
  Week 12 | 3240 (916)

6. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of DFV890
Description: AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast). DFV890 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8). DFV890 was determined by a validated LC-MS/MS method; the lower limit of quantification (LLOQ) is 1 ng/mL.
Time Frame: Week 2 and Week 12: pre-dose, 1h, 3h, 5h, 8h
Population: The PK analysis set included all participants with at least 1 available valid (i.e., not flagged for exclusion) PK concentration measurement, who received DFV890 and with no protocol deviations that impact on PK data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | DFV890
Number analyzed (Participants) | 52
h*ng/mL
  Week 2 | 9070 (3940)
  Week 12: number analyzed (Participants) | 50
  Week 12 | 19300 (6370)

7. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to 12 Hours (AUC0-12h) of DFV890
Description: AUC(0-12h) is the area under the plasma concentration-time curve from time zero to 12 hours. To calculate AUC0-12h (corresponding to AUCtau, or AUC within a dosing interval), the concentration at 0 hours was used also as a 12 hours time point or, if not feasible, AUC0-12h was extrapolated. DFV890 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8). DFV890 was determined by a validated LC-MS/MS method; the lower limit of quantification (LLOQ) is 1 ng/mL.
Time Frame: Week 2 and Week 12: pre-dose, 1h, 3h, 5h, 8h
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | DFV890
Number analyzed (Participants) | 47
h*ng/mL
  Week 2 | 12300 (5120)
  Week 12: number analyzed (Participants) | 45
  Week 12 | 26700 (8210)

8. Secondary Outcome: Pre-dose Trough Concentration (Ctrough) of DFV890
Description: DFV890 plasma concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8). DFV890 was determined by a validated LC-MS/MS method; the anticipated lower limit of quantification (LLOQ) is 1 ng/mL.
Time Frame: Week 2 and Week 12: pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DFV890
Number analyzed (Participants) | 55
ng/mL
  Week 2 | 653 (360)
  Week 12: number analyzed (Participants) | 51
  Week 12 | 1530 (665)

9. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Other Symptoms Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is other symptoms (eg., stiffness, swelling, clicking) consisting of 7 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Change from baseline in other symptoms score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | 6.9 (1.94) | 2.0 (2.09)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | 12.3 (2.25) | 8.1 (2.31)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | 16.2 (2.55) | 12.6 (2.59)
  Week 12: number analyzed (Participants) | 45 | 41
  Week 12 | 19.3 (2.57) | 13.8 (2.67)

10. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the Function in Daily Living consisting of 17 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no impact on function in daily living and 0 indicating extreme impact on function in daily living) is calculated for each subscale. Change from baseline in KOOS daily living function score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | 5.7 (1.71) | 6.9 (1.85)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | 12.7 (1.92) | 12.0 (1.98)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | 17.2 (2.40) | 15.8 (2.46)
  Week 12: number analyzed (Participants) | 45 | 41
  Week 12 | 21.1 (2.46) | 19.4 (2.57)

11. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Sport and Recreation Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the function in sport and recreation consisting of 5 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no impact on sport and recreation and 0 indicating extreme impact on sport and recreation) is calculated for each subscale. Change from baseline in function in sport and recreation score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | 3.1 (2.40) | 7.5 (2.60)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | 11.8 (2.71) | 10.7 (2.79)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | 17.7 (3.37) | 14.4 (3.43)
  Week 12: number analyzed (Participants) | 45 | 41
  Week 12 | 16.6 (3.30) | 19.3 (3.41)

12. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Knee-related Quality of Life (QOL) Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the knee-related quality of life consisting of 4 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no impact on knee-related quality of life and 0 indicating extreme impact on knee-related quality of life) is calculated for each subscale. Change from baseline in knee related quality of life score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | 5.0 (1.80) | 6.3 (1.93)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | 13.2 (2.19) | 11.7 (2.26)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | 17.1 (2.54) | 13.2 (2.58)
  Week 12: number analyzed (Participants) | 45 | 41
  Week 12 | 18.4 (2.65) | 16.3 (2.75)

13. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is pain frequency/severity during functional activities consisting of 9 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no pain and 0 indicating extreme pain) is calculated for each subscale. Change from baseline in KOOS pain score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Week 2, 4, 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | 7.8 (1.78) | 6.9 (1.92)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | 14.8 (1.92) | 11.4 (1.98)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | 19 (2.47) | 13.3 (2.51)

14. Secondary Outcome: Change From Baseline in Numeric Rating Scale (NRS) for Pain
Description: The Numerical Rating Scale (NRS) Pain is a subjective assessment in which individuals rate their pain on an eleven-point numerical scale. NRS pain score ranges from 0-10 and for analyses were transformed to a 0-100 scale to be consistent with KOOS pain scores. A negative change from baseline implied improvement in pain. The NRS Pain instrument had a recall period of 24 hours and the participants were asked to rate the pain intensity at its worst. Change from baseline in NRS pain score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint, baseline-by-timepoints interaction and treatment-by-timepoints interaction as fixed effects. Missing data is assumed to be Missing at Random (MAR).
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 47 | 43
score on scale
  Week 2: number analyzed (Participants) | 47 | 39
  Week 2 | -10.5 (2.43) | -11.5 (2.6)
  Week 4: number analyzed (Participants) | 45 | 42
  Week 4 | -18.1 (2.65) | -14.4 (2.74)
  Week 8: number analyzed (Participants) | 44 | 43
  Week 8 | -27.2 (2.86) | -18.8 (2.92)
  Week 12: number analyzed (Participants) | 45 | 41
  Week 12 | -29.7 (3.07) | -23.9 (3.19)

15. Post Hoc Outcome: Number of Participants With Neutrophil Counts <2.03 x 10⁹/l (Lower Limit of Normal)
Description: Neutrophils, a type of white blood cell essential for fighting infection, are measured in blood samples. Instances of neutrophil counts falling below the lower limit of normal were not consistently reported by all Principal Investigators as Adverse Events. To address this, an ad-hoc outcome measure was introduced to capture 'Neutrophil counts below the lower limit' based on laboratory data.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, End of Study (up to approximately 14 weeks)
Population: Safety analysis set: All randomized participants that have received any study drug and had a valid measurement at the respective time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | DFV890 | Placebo
Number analyzed (Participants) | 58 | 57
Participants
  Baseline | 3 | 1
  Week 2: number analyzed (Participants) | 52 | 56
  Week 2 | 11 | 1
  Week 4: number analyzed (Participants) | 51 | 52
  Week 4 | 12 | 1
  Week 8: number analyzed (Participants) | 51 | 55
  Week 8 | 9 | 0
  Week 12: number analyzed (Participants) | 50 | 51
  Week 12 | 15 | 2
  End of Study: number analyzed (Participants) | 53 | 53
  End of Study | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 114 days.
Groups:
- DFV890 10mg: DFV890 was administered orally twice per day, 10 mg during 2 weeks. AEs that started while on DFV890 10 mg (week 1 and 2).
- DFV890 25mg: DFV890 was administered orally twice per day, 10 mg during 2 weeks and 25 mg during the next 10 weeks. AEs that started while on DFV890 25 mg (weeks 3 to 12 + 30 days follow up).
- Total: Total
Arm/Group | DFV890 10mg | DFV890 25mg | DFV890 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/57 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/58 | 1/58 | 1/57 | 2/115
Other Adverse Events (participants affected / at risk) | 3/58 | 19/58 | 20/58 | 11/57 | 31/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DFV890 10mg (N=58) | DFV890 25mg (N=58) | DFV890 (N=58) | Placebo (N=57) | Total (N=115)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFV890 10mg (N=58) | DFV890 25mg (N=58) | DFV890 (N=58) | Placebo (N=57) | Total (N=115)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 5
COVID-19 (Infections and infestations) | 0 | 5 | 5 | 2 | 7
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3 | 4 | 7
Neutrophil count decreased (Investigations) | 0 | 10 | 10 | 2 | 12
Headache (Nervous system disorders) | 1 | 3 | 4 | 3 | 7

LIMITATIONS AND CAVEATS:
Due to MedDRA version 27.1, the reported term 'interstitial pneumonia' was decoded to the Preferred Term 'interstitial lung disease' in the Adverse Events report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT04886258/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04886258/SAP_001.pdf